CLINICAL TRIAL: NCT03106168
Title: Evaluation of Anesthetic Efficacy in Extraction on Mandibular Molars With Periapical Granuloma
Brief Title: Evaluation of Anesthetic Efficacy in Extraction on Mandibular Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Klouczek Carrocini, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Extraction
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-06

CONDITIONS: Local Anesthetics; Tooth Extraction
Keywords: Extraction; Local Anesthetic; Mepivacaine; Mandibular Molar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With periapical granuloma (Experimental): Patients presenting periapical granuloma in mandibular molar teeth, diagnosed by periapical radiography
  Interventions: Procedure: Extraction of mandibular molar
- Without periapical granuloma (Experimental): Patients without periapical granuloma in mandibular molar teeth, diagnosed by periapical radiography
  Interventions: Procedure: Extraction of mandibular molar

INTERVENTIONS:
Procedure: Extraction of mandibular molar — Patients who require extraction of mandibular molars will be submitted to surgery

SUMMARY:
To evaluate subjectively and objectively the quality and efficacy of local anesthetic block with mepivacaine in simple extraction of mandibular molar. Provide and collect information such as: signs and symptoms, quality of anesthetic block, quantify pain and / or discomfort, as well as medication used, both preoperatively and postoperatively.

DETAILED DESCRIPTION:
Anamnesis and clinical diagnosis of patients, with indication of extraction, will be performed by the Emergency Department of the School of Dentistry of the University of São Paulo (SDUSP). Of these, 80 patients with mandibular molar teeth extraction, with and without apparent apical lesion radiographically identified in the initial imaging examination will be included. They must be over 16 years old, with good judgment and good general health, who have availability of return to the clinic for postoperative follow-up and aware of the Term of Consent.

After the anamnesis, clinical and radiographic examinations for diagnosis and inclusion in the study, they will receive information on the procedure to be submitted, mainly on the quality of the local anesthetic block, quantification of pain and / or discomfort, and what will occur on the days after the procedure, such as guidelines and post-operative care (PO).

The clinical procedure (extraction) will follow the protocol of attendance of the Emergency Department of SDUSP, which is consistent with the surgical practice in force in this School and in other Dentistry Schools. In clinical care, patients will be questioned about the presence of discomfort and / or pain, indicated on the visual analogue scale (VAS score 0, score 1, score 2 or pain score 3). They will be informed about the effects of anesthesia, the use of the pulptest sensitivity test, absence of sensitivity in soft tissue and pulp after anesthesia, and the need for complementation with more local anesthetic (Mepivacaine and Noradrenaline) and / or incorporation of other anesthetic techniques.

To obtain basal tooth responsiveness patterns, prior to anesthesia, the pulptest will be applied to vital teeth of the quadrant that will receive intervention. The same will be reapplied after the injection of the anesthetic, in order to verify the installation of the blockade. Only after the anesthetic blockade has been confirmed and installed, both pulp ("Pulptest"), and soft tissues, the patient will be included in the research, initiating the surgical procedure. Any discomfort or complaint that the patient may have during the transoperatory period will be considered and, if necessary, we will use anesthetic complementation, which is recorded. In the postoperative period, these patients will have the opportunity to report some discomfort and pain, through a questionnaire, which will be filled and returned on the day of removal of suture, as well as intercurrence and / or need to use the suggested medication in case of pain.

The information obtained in this study will be inserted in Excel spreadsheet for descriptive analysis, statistics and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients that need extraction of one or more dental elements, older than or equal to sixteen and less than sixty, will be included, obligatorily with local surgical and systemic need and opportunity. They should be literate, able to read and understand, with discernment and able to answer the survey questionnaire. The indication for extraction should be attributed to caries destruction, periodontal impairment, large trauma damage, root fractures, orthodontic indication, prosthetic / rehabilitative or presence of residual roots.

Exclusion Criteria:

* Patients over sixty, smokers, pregnant women, immunosuppressed, users of steroids, antidepressive and / or other psychiatric medications, users of illicit drugs, carriers of hemorrhagic disorders, with previous history of radiotherapy in the oral cavity, patients with metabolic and / or glandular bone disorders of chronic renal failure. Patients in whom the initial anesthesia does not install after a tube, without analgesia of part of the lip and tongue, or without numerical alteration in the pulp test, will also be excluded, characterizing failure in the anesthetic technique.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Anesthetic efficacy | 10 minutes after anesthetic technique
  The anesthetic efficacy will be analyzed through the use of a verbal numerical scale used during the pulpectomy procedure

SECONDARY OUTCOMES:
Pulpal Anesthesia | 10 minutes after anesthetic technique
  Pulp anesthesia was defined as the absence of a positive response to the Pulptest after 10 minutes of the inferior alveolar nerve block in the teeth adjacent to the one selected for extraction
Postoperative pain | seven days after the extraction
  A postoperative evaluation of pain and discomfort was carried out by the patient in the first seven days after the surgery through the analysis of a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bruno k Carrocini, Ms, Principal Investigator — University of Sao Paulo
Locations (1):
- Serviço de Urgência da Faculdade de Odontologia de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided